CLINICAL TRIAL: NCT04932512
Title: An Adaptive Two-Part Phase 2, Multi-Center, Randomized, Double Blind, Placebo-Controlled Study to Assess the Safety, Efficacy, and Pharmacokinetics of Multiple Doses of ION224 Administered Once Monthly in Adult Subjects With Confirmed Non-Alcoholic Steatohepatitis
Brief Title: A Study to Assess the Safety, Efficacy, and Pharmacokinetics of Multiple Doses of ION224
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION224-CS2
Record Dates: First submitted 2021-06-10; First posted 2021-06-21 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Steatohepatitis, Nonalcoholic
Keywords: Non-Alcoholic Steatohepatitis; Non-alcoholic Fatty Liver Disease Activity Score; Alanine Aminotransferase; Aspartate Aminotransferase
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ION224 (Experimental): Multiple doses of ION224 will be administered by SC injection once every 4 weeks for up to 49 weeks.
  Interventions: Drug: ION224
- Placebo (Placebo Comparator): Multiple doses of matching placebo will be administered by SC injection once every 4 weeks for up to 49 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ION224 — ION224 will be administered by SC injection.
  Arms: ION224
Other: Placebo — ION224-matching placebo solution will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of multiple ION224 doses when administered by subcutaneous (SC) injection for 49 weeks (end of the treatment [EOT]) on non-alcoholic steatohepatitis (NASH) histologic improvement and to assess the effect on liver steatosis by magnetic resonance imaging-determined proton density fat fraction (MRI-PDFF), additional changes in NASH histologic features, liver biochemistry tests, and plasma lipid profile.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, randomized, placebo-controlled study of ION224 in up to 150 participants. The study consists of 3 periods: 1) Screening Period: Week -8 to Week -1 (up to 8 weeks); 2) Treatment Period up to Week 49; and 3) Post-Treatment Period: Week 50 to Week 62 (12 weeks).

Initially, 48 patients will be enrolled in three different dose cohorts to receive ION224 or placebo every four weeks and based on safety and effects on liver steatosis (assessed at Week 15), two dose cohorts will be selected to be expanded. After dose selection, an additional 102 patients will be enrolled in the 2 selected dose cohorts and will receive ION224 or placebo for up to 49 weeks. Participants in the 3rd cohort (not selected) will continue to complete up to 49 weeks of treatment without any cohort expansion.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than or equal to (≥) 18 and less than or equal to (≤) 75 years old at the time of informed consent
* Body mass index ≥ 25 kg/m^2 and ≥ 22 kg/m^2 for participants of Asian race, as assessed during screening
* Liver fat ≥ 10% as assessed by MRI-PDFF before randomization
* Presence of NASH confirmed by centrally read liver biopsy
* Weight loss < 5% after historical biopsy. Otherwise, weight loss < 5% in the previous 3 months prior to randomization
* ALT and AST ≤ 200 units per liter (U/L) and confirmed to be stable
* Total Bilirubin ≤ 1.3 milligrams per deciliter (mg/dL) and confirmed to be stable

Exclusion Criteria:

* Prior or planned (during the Study Period) bariatric surgery or previous bariatric surgery within 2 years prior to screening
* History of solid organ transplant
* Screening laboratory values that would render a participant unsuitable for inclusion, including but not limited to:

  * Clinically significant albuminuria or proteinuria
  * Positive test for blood on urinalysis
  * Estimated glomerular filtration rate (eGFR) < 60 milliliters (mL)/minute (min)/1.73 square meter (m^2)
  * Hemoglobin A1c (HbA1c) > 9.5%
  * Platelet count < 170 × 10^9/liter (L)
* Diagnosis of Gilbert's syndrome
* Known history of or evidence of liver disease other than NASH
* Clinical evidence of liver decompensation
* Active SARS-CoV-2 infection (COVID-19) or confirmed SARS-CoV-2 infection-related complication within 8 weeks of Screening
* Uncontrolled arterial hypertension
* History of bleeding diathesis or coagulopathy
* Participants with known intolerance to magnetic resonance imaging (MRI) or with conditions contraindicated for MRI Procedures
* History of, or current hard drug or alcohol abuse within 2 years prior to Screening
* Use of drugs historically associated with NAFLD for more than 2 weeks in the year prior to Screening
* Use of obeticholic acid, ursodeoxycholic acid, icosapent ethyl, niacin, PCSK9 inhibitors, and bile acid sequestrants
* Participants taking the following medicines UNLESS on a stable dose:

  * Anti-diabetic medications
  * statins, fenofibrate, and ezetimibe
  * Estrogen containing contraceptives
  * Glucagon-like peptide (GLP)-1 agonists
  * Pioglitazone
  * Vitamin E at doses ≤ 800 international unit (IU)/day
  * Herbal medicines, other prescription medicines, vitamins or supplements known to affect lipid metabolism
* Other protocol-defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With at Least 2-point Reduction in Non-alcoholic Fatty Liver Disease Activity Score (NAS) With at least 1-point Improvement in Hepatocellular Ballooning or Lobular Inflammation, and Without Worsening in Fibrosis Stage at EOT | Up to Week 49
  The NAS is a histology grading score composed on the assessment of steatosis (scale 0-3), hepatocellular ballooning (scale 0-2), and lobular inflammation (scale 0-3), with higher scores indicating more severe hepatitis. Worsening of fibrosis is defined as an increase in fibrosis of at least one stage on the Kleiner fibrosis classification: fibrosis stages range from 0-4, with higher scores indicating greater fibrosis (0=None, 4=Cirrhosis).

SECONDARY OUTCOMES:
Change From Baseline in Hepatic Fat Content Measurement as Evaluated by MRI-PDFF and Calculated by an Independent, Blinded-To-Treatment, Central Reader | Baseline up to Week 15, Week 29 and Week 49
Percentage of Participants Achieving Non-alcoholic Steatohepatitis (NASH) Resolution, as Defined by Scores of 0 for Ballooning and 0 or 1 for Inflammation by the NAS, and Without Worsening of Fibrosis, Assessed Through Liver Biopsy at the EOT | Up to Week 49
Percentage of Participants Achieving Reduction of at Least 1 Stage in the Fibrosis Score, and Without Worsening of Steatohepatitis by the NAS, Assessed Through Liver Biopsy at the EOT | Up to Week 49
Percentage of Participants Achieving a Combination of NASH Resolution and a 1 Stage Improvement in Fibrosis at the EOT | Up to Week 49
Percentage of Participants With Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) Less than or Equal to (≤) 1.5 Upper Limit of Normal (ULN) at the EOT | Up to Week 49
Absolute Change From Baseline in Liver-related Laboratory Test - ALT | Baseline up to Week 49
Absolute Change From Baseline in Liver-related Laboratory Test - AST | Baseline up to Week 49
Absolute Change From Baseline in Liver-related Laboratory Test - Total Bilirubin | Baseline up to Week 49
Absolute Change From Baseline in Liver-related Laboratory Test - Gamma-glutamyl Transferase | Baseline up to Week 49
Absolute Change From Baseline in Plasma Fasting Lipid Profile Test - Triglyceride (TG) | Baseline up to Week 49
Absolute Change From Baseline in Plasma Fasting Lipid Profile Test - Total Cholesterol | Baseline up to Week 49
Absolute Change From Baseline in Plasma Fasting Lipid Profile Test - Low-density Lipoprotein-cholesterol (LDL-c) | Baseline up to Week 49
Absolute Change From Baseline in Plasma Fasting Lipid Profile Test - High-density Lipoprotein-cholesterol (HDL-c) | Baseline up to Week 49
Maximum Observed Plasma Concentration (Cmax) of ION224 and Metabolites | Baseline up to Week 49
Time to Cmax (Tmax) of ION224 and Metabolites | Baseline up to Week 49
Area Under the Plasma Concentration-time Curve (AUC) of ION224 and Metabolites | Baseline up to Week 49
Plasma Half-life (t½) of ION224 and Metabolites | Baseline up to Week 49

CONTACTS AND LOCATIONS:
Locations (51):
- United States (50):
  - Arizona Liver Health-Chandler, Chandler, Arizona
  - Arizona Liver Health, Glendale, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Arkansas Gastroenterology - North Little Rock, North Little Rock, Arkansas
  - GW Research, Inc., Chula Vista, California
  - National Research Institute - Gardena, Gardena, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - National Research Institute Panorama City, Panorama City, California
  - National Research Institute - Santa Ana, Santa Ana, California
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Southwest General Medical Center, Fort Myers, Florida
  - Evolution Clinical Trials, INC, Hialeah Gardens, Florida
  - ClinCloud, LLC., Maitland, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - La Salud Research, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Floridian Clinical Research, LLC., Miami Lakes, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Tandem Clinical Research GI, Houma, Louisiana
  - Tandem Clinical Research GI, LLC., Marrero, Louisiana
  - Tandem Clinical Research GI, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Advanced Research Institute, Reno, Nevada
  - Clarity Clinical Research, East Syracuse, New York
  - Tandem Clinical Research GI, LLC., New York, New York
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Aventiv Research, Inc., Columbus, Ohio
  - Clinical Research Institute of Ohio, Westlake, Ohio
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Pinnacle Clinical Research, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Velocity Clinical Research, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - R&H Clinical Research, Inc., Katy, Texas
  - DHR Health Institute for Research and Development, McAllen, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - Granger Medical Clinic, Riverton, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loomba R, Morgan E, Yousefi K, Li D, Geary R, Bhanot S, Alkhouri N; ION224-CS2 Investigators. Antisense oligonucleotide DGAT-2 inhibitor, ION224, for metabolic dysfunction-associated steatohepatitis (ION224-CS2): results of a 51-week, multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2025 Aug 23;406(10505):821-831. doi: 10.1016/S0140-6736(25)00979-1. PMID 40849139